CLINICAL TRIAL: NCT07273435
Title: Comparison of Predicted and Achieved Crown Movements in Adult Spacing Cases Treated With 3D Direct-printed Aligners: A Prospective Clinical Trial
Brief Title: Crown Movement in Cases Treated With Direct Printed Aligners
Acronym: DPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Collaborators: Beni-Suef University (Other); British University In Egypt (Other)
Responsible Party: Principal Investigator, rim fathalla, Rim Mohamed Fathalla Eissa, Suez Canal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #REC-FDBSU/06032025-02/AR
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Effect of Direct Printed Aligners on Crown Movement
Keywords: Direct printed aligners crown movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with spacing (Experimental): Patients will receive direct printed aligners to treat the spacing
  Interventions: Other: Direct printed aligners

INTERVENTIONS:
Other: Direct printed aligners — Direct printed aligners After intraoral scanning, patients will receive Direct printed aligners, each set will be changed after 10 days, till the patients finish their treatment, then a post intraoral scan will be taken from each patient.

SUMMARY:
This study aims to evaluate the efficiency of direct 3D printed aligners in achieving the crown movement of upper and lower incisors in patients with spacing during space closure and to compare them with the predicted tooth movements

DETAILED DESCRIPTION:
This study will be carried out on 23 patients seeking orthodontic treatment at the outpatient orthodontic clinics at the Faculty of Dentistry, Suez Canal, Beni Suef, and British Universities.

The inclusion criteria are: patients aged 18-45 years, with full permanent dentition (excluding third molars), generalized spacing or spacing between anterior teeth, normal skeletal relationships, and Angle Class I or mild Class II malocclusions. Patients with the following criteria will be excluded: patients with missing or extracted permanent teeth (excluding third molars), periodontally compromised teeth, who need any form of hybrid orthodontic treatment (a fixed appliance with aligners), any signs or symptoms of temporomandibular disorders, severe Angle Class II or Class III malocclusions, crowding, and Class II or Class III skeletal discrepancy.

Methods:

1. Intraoral scans will be obtained for the upper and lower arches followed by a 3D simulation before treatment to check the biomechanics and movements of the treatment.
2. After setting up the 3D digital design for treatment, we will begin the fabrication of 3D printed aligners.
3. The patient will be instructed to use the aligner, and instructions will be given to the patient to put aligners in warm water before wearing them. This activates their shape memory allowing them to fit more easily and comfortably, thus reducing stress on the aligners.
4. The Patient will change the aligners every week according to the manufacturer's instructions and at the end of treatment, a new 3D scanning for the patient's dental arches will be taken to obtain the actual model after treatment.
5. The virtual pre-treatment model obtained before, and the actual post-treatment model will be exported as STL files and imported into digital software as virtual pre-treatment and actual post-treatment models.
6. The virtual pre-treatment, virtual and achieved post-treatment models will be superimposed digitally.
7. After superimposition, a 3D coordinate system will be generated for tooth movement measurements. After determining the reference points on the pre-treatment model, they will be transferred onto actual and virtual post-treatment models through tooth crown surface superimposition. The achieved and predicted changes in crown movement of the upper and lower incisors will be calculated.

All numerical data will be collected for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18- 45 years old.
* Non- extraction treatment.
* Angle Class I or Class II dental malocclusion with generalized or localized anterior spacing.
* Normal probing depth.

Exclusion Criteria:

* Active periodontal disease.
* Crowding cases.
* Systemic diseases or medications that alter bone metabolism or tooth movement.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of direct 3D printed aligners in achieving the planned crown movement of upper and lower incisors ( measured in mm). | 9-12 months
  Compare the achieved crown movements with the predicted crown movements of the upper and lower incisors in spacing cases treated with Directed printed aligners by comparing the pre virtual set up with post treatment set up of the cases using superimposition digital software.

CONTACTS AND LOCATIONS:
Overall Officials: Rim M Fathalla, PhD of Orthodontics, Principal Investigator — Suez Canal University
Locations (3):
- Egypt (3):
  - Beni-Suef University, Banī Suwayf
  - British University in Egypt, Cairo
  - Suez Canal University, Ismailia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hertan E, McCray J, Bankhead B, Kim KB. Force profile assessment of direct-printed aligners versus thermoformed aligners and the effects of non-engaged surface patterns. Prog Orthod. 2022 Nov 29;23(1):49. doi: 10.1186/s40510-022-00443-2. PMID 36443390
- [Result] Lee SY, Kim H, Kim HJ, Chung CJ, Choi YJ, Kim SJ, Cha JY. Thermo-mechanical properties of 3D printed photocurable shape memory resin for clear aligners. Sci Rep. 2022 Apr 15;12(1):6246. doi: 10.1038/s41598-022-09831-4. PMID 35428796
- [Result] McKay A, McCray J, Bankhead B, Lee MM, Miranda G, Adel SM, Kim KB. Forces and moments generated during extrusion of a maxillary central incisor with clear aligners: an in vitro study. BMC Oral Health. 2023 Jul 17;23(1):495. doi: 10.1186/s12903-023-03136-2. PMID 37461004
- [Result] Kravitz ND, Kusnoto B, Agran B, Viana G. Influence of attachments and interproximal reduction on the accuracy of canine rotation with Invisalign. A prospective clinical study. Angle Orthod. 2008 Jul;78(4):682-7. doi: 10.2319/0003-3219(2008)078[0682:IOAAIR]2.0.CO;2. PMID 18302468
- [Result] Weir T. Clear aligners in orthodontic treatment. Aust Dent J. 2017 Mar;62 Suppl 1:58-62. doi: 10.1111/adj.12480. PMID 28297094